CLINICAL TRIAL: NCT04942093
Title: NUTritional Impact of a Hypocaloric Hyperprotein Diet Before Obesity Surgery
Acronym: NUTRACOB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/0414/HP
Record Dates: First submitted 2021-06-11; First posted 2021-06-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Diet, Healthy; Obesity, Visceral; Bariatric Surgery Candidate
Keywords: diet; obesity; bariatric surgery
MeSH Terms: conditions — Obesity, Abdominal; Obesity | interventions — Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With diet (Experimental): A low-calorie, high-protein diet will be prescribed to the patient for a period of 4 weeks. The diet will be done the 4 weeks before the bariatric surgery
  Interventions: Dietary Supplement: With low-calorie, high-protein diet
- Without diet (Other): A low-calorie, high-protein diet will not be prescribed to the patient for a period of 4 weeks.
  Interventions: Dietary Supplement: Without low-calorie, high-protein diet

INTERVENTIONS:
Dietary Supplement: With low-calorie, high-protein diet — A low-calorie, high-protein diet will be prescribed to the patient for a period of 4 weeks. The diet will be done the 4 weeks before the bariatric surgery
  Arms: With diet
Dietary Supplement: Without low-calorie, high-protein diet — A low-calorie, high-protein diet will not be prescribed to the patient for a period of 4 weeks.
  Arms: Without diet

SUMMARY:
Obesity is a major public health problem and is constantly on the rise. Therapeutic approaches based on dietary advice, physical activity and the management of psychological difficulties are not always sufficient to achieve a lasting weight reduction.

Bariatric surgery (or obesity surgery), accompanied by therapeutic education and adequate medical and dietary monitoring, can lead to significant and lasting weight loss. It is indicated as a second-line treatment for patients who have failed medical treatment, whose BMI is greater than or equal to 40 or whose BMI is greater than or equal to 35 with comorbidities (type 2 diabetes, arterial hypertension, obstructive sleep apnoea-hypopnoea syndrome, severe joint disorders).

The surgeon may be very bothered by the intra-abdominal fat mass and especially by steatotic hepatomegaly (increase in the size of the liver and its fat load).

Faced with this problem, various preoperative strategies such as the placement of an intra gastric balloon have been tried to decrease the size of the liver but a systematic review from 2016 indicates that a low calorie diet is preferable. Preoperative weight loss can reduce fat load and liver volume very rapidly. This meta-analysis shows that all low-calorie, high-protein diets are effective and that the optimal duration (4 weeks), compliance and tolerance are important factors for success.

DETAILED DESCRIPTION:
Obesity is a major public health problem and is constantly on the rise. Therapeutic approaches based on dietary advice, physical activity and the management of psychological difficulties are not always sufficient to achieve a lasting weight reduction.

Bariatric surgery (or obesity surgery), accompanied by therapeutic education and adequate medical and dietary monitoring, can lead to significant and lasting weight loss. It is indicated as a second-line treatment for patients who have failed medical treatment, whose BMI is greater than or equal to 40 or whose BMI is greater than or equal to 35 with comorbidities (type 2 diabetes, arterial hypertension, obstructive sleep apnoea-hypopnoea syndrome, severe joint disorders).

The surgeon may be very bothered by the intra-abdominal fat mass and especially by steatotic hepatomegaly (increase in the size of the liver and its fat load).

Faced with this problem, various preoperative strategies such as the placement of an intra gastric balloon have been tried to decrease the size of the liver but a systematic review from 2016 indicates that a low calorie diet is preferable. Preoperative weight loss can reduce fat load and liver volume very rapidly. This meta-analysis shows that all low-calorie, high-protein diets are effective and that the optimal duration (4 weeks), compliance and tolerance are important factors for success.

However, there is no consensus on the benefit/risk balance of a preoperative diet and there is considerable variability in approach at national and international level.

The present clinical study involves a triad of dietician, surgeon, physician (endocrinologist/nutritionist or internist) to secure this diet. It could provide a database to help estimate the risk of undernutrition in the obese subject.

This diet, designed to facilitate the surgical procedure and potentially reduce intraoperative complications, is inexpensive, easily accessible and reproducible by other teams. This innovative management could standardise the preoperative management of patients undergoing bariatric surgery at national level. It would also improve the results of bariatric surgery both in the short term by reducing complications and in the long term by increasing weight reduction as reported in the Livhits meta-analysis. The risk of undernutrition should be reduced by this hypocaloric hyperprotein diet and consequently cancel out the increased risk of mortality, infections, delayed healing, longer hospital stay and the costs that this would entail.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for bariatric surgery (according to HAS criteria) whose sleeve gastrectomy is scheduled
* Patient with morbid obesity (BMI ≥ 40)
* Age ≥ 18 years and ≤ 65 years
* Haemoglobinemia ≥ 12 g/dL in men and ≥ 11 g/dL in women
* Patient speaking and understanding French
* Adult having read and understood the information letter and signed the consent form
* Woman of childbearing age with effective / very effective contraception (Cf. CTFG) (estrogen-progestin or intrauterine device or tubal ligation) prior to surgery and a negative -HCG blood pregnancy test at inclusion, for the duration of the study
* Postmenopausal woman: confirmatory diagnosis (non-medically induced amenorrhoea for at least 12 months prior to the inclusion visit)
* Patient affiliated with, or beneficiary of a social security (health insurance) category

Exclusion Criteria:

* Contraindication to bariatric surgery detected during the preoperative assessment
* Medical contraindication to a restrictive diet
* Type I or II insulin-requiring diabetes
* Severe renal insufficiency defined by a blood filtration rate < 30 mL/min
* Person wearing a pacemaker or any other implant with the same functions (cochlear implant, bladder battery, etc.)
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection / sub-guardianship or curatorship
* A history of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol or to prevent him/her from giving informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Poor diet tolerance | 4 weeks after the beggining of the diet
  At least one of the following biological abnormalities at the end of the diet period:
  * Lymphopenia acquired during the diet
  * Anemia (Hb<11g/dL for men Hb<10g/dL for women) or a decrease in hemoglobin of more than 2 g/dL
  * Onset or worsening of vitamin B1 deficiency from baseline (Vit B1 < 78 nmol/L)
  OR
  At least one of the following clinical abnormalities:
  * Decrease in muscle strength (difference in muscle strength measured with a HandGrip at Visit 2 and Visit 3) greater than three standard deviations from the matched Visit 3 - visit 2 differences of the control group after removal of measurement bias on a log-transformed strength variable, associated with weight loss > 5% in 1 month or a decrease in percent lean mass ≥ 1% relative to visit 2
  * Any permanent discontinuation

SECONDARY OUTCOMES:
Weight loss | 4 weeks after the beggining of the diet and 3 months postoperatively
  Weight difference between Visit 3 and Visit 2
Reduced muscle strength | 4 weeks after the beggining of the diet
  Difference in muscle strength measured with a HandGrip at Visit 2 and Visit 3)
Comparison of the quality of life between "with diet" and "without diet" with "EQVOD" questionnaire | Baseline, 4 weeks after the beggining of the diet and 3 months postoperatively
  Evaluated using the EQVOD questionnaire at baseline (V2), end of diet (V3) and 3 months postoperatively Score from 36 to 180
Evolution of physical activity | Baseline, 4 weeks after the beggining of the diet and 3 months postoperatively
  Physical activity evaluated using the Ricci et Gagnon questionnaire at baseline (V2), end of diet (V3) and 3 months postoperatively
Digestive tolerance | during the 4 weeks of the diet
  Digestive tolerance evaluated using auto-questionnaire about nausea, vomiting, diarrhoea, constipation forthe interventional group, in the month of the diet
Compliance | during the 4 weeks of the diet
  Evaluated by a food diary and the full bottles (not consumed) brought back for the intervention group, in the month of the diet
Degree of exposure | one day from surgery
  Assessment of the degree of exposure of the oesogastric junction and hepatomegaly on a subjective scale of 1 to 5 by the surgeon
Operating time | one day from surgery
  Number of hours and minuts about surgery
Length of hospital stay | Four months from surgery
  Number of days in hospital for the surgery
Intraoperative and postoperative complications | Between surgery and 3 months postoperatively
  Delayed healing, infection and cancellation of surgery or conversion to laparotomy) up to 3 months post-operatively

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Ch Dieppe, Dieppe
  - HPE, Le Havre
  - CHU de ROUEN, Rouen

IPD SHARING:
Plan to Share IPD: No